CLINICAL TRIAL: NCT02438306
Title: Randomized Controlled Pivotal Trial of Autologous Bone Marrow Mononuclear Cells Using the CardiAMP Cell Therapy System in Patients With Ischemic Heart Failure (CardiAMP Heart Failure Trial)
Brief Title: CardiAMP™ Cell Therapy for Heart Failure Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioCardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-14-001
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- CardiAMP cell therapy (Experimental): Placement of an introducer guidewire, performance of a left ventriculogram, and treatment with autologous cell therapy.
  Interventions: Biological: Autologous cell therapy
- Sham Comparator (Sham Comparator): Placement of an introducer guidewire and performance of a left ventriculogram with no autologous cell therapy treatment.
  Interventions: Other: Sham

INTERVENTIONS:
Biological: Autologous cell therapy — Autologous cell therapy delivered into the heart muscle using the CardiAMP Cell Therapy System. The CardiAMP Cell Therapy System consists of the CardiAMP Cell Separator, a cardiac delivery catheter, and flexible tip guide catheter.
  Arms: CardiAMP cell therapy
Other: Sham — An introducer guidewire is placed into the heart and left ventriculography is performed just like it is in the Experimental Arm but no autologous cell therapy is delivered.
  Arms: Sham Comparator

SUMMARY:
This is a prospective, multi-center, randomized, controlled, patient- and evaluator-blinded study comparing treatment with the CardiAMP cell therapy to a sham control treatment. A roll-in phase with a maximum of 10 subjects may occur.

DETAILED DESCRIPTION:
Heart failure is a clinical condition in which the output of blood from the heart is insufficient to meet the metabolic demands of the body. In 2015, the American Heart Association, or AHA, report on heart disease statistics estimated that there are 5.7 million Americans over the age of 20 that have heart failure. Heart failure is increasingly prevalent due to the aging population and the increase in major cardiovascular risk factors, including obesity and diabetes.

The AHA also estimates that one in five adults will develop heart failure after the age of 40. During heart failure progression, the heart steadily loses its ability to respond to increased metabolic demand, and mild exercise soon exceeds the heart's ability to maintain adequate output. Towards the end stage of the disease, the heart cannot pump enough blood to meet the body's needs at rest. At this stage, fluids accumulate in the extremities or in the lungs making the patient bedridden and unable to perform the activities of daily living. The long-term prognosis associated with heart failure is approximately 50% mortality at five years following the initial diagnosis.

CardiAMP cell therapy is a comprehensive therapeutic treatment that comprises (i) a point of care cell processing platform and (ii) a biotherapeutic delivery system. CardiAMP cell therapy is the first comprehensive therapeutic treatment utilizing a patient's own cells for the treatment of ischemic heart failure with reduced ejection fraction. In the screening process, the physician extracts a small sample of the patient's bone marrow in an outpatient procedure performed under local anesthesia. The clinic sends the sample to a central diagnostic lab, which tests the sample. For the study treatment, a clinician collects and then prepares the patient's own bone marrow mononuclear cells, or autologous cells, using the CardiAMP point of care cell processing platform, which a cardiologist then delivers into the heart using the Helix biotherapeutic delivery system.

BioCardia intends to submit data obtained from this clinical trial in a Pre-Market Approval Application to the United States Food and Drug Administration

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) Class II or III
* A diagnosis of chronic ischemic left ventricular dysfunction secondary to myocardial infarction (MI) as defined by selected criteria.
* On stable evidence-based medical and device therapy for ischemic etiology heart failure, per the ACC/AHA Heart Failure guidelines, for at least three (3) months prior to randomization.
* Left ventricular ejection fraction between 20% and 40%.
* Qualification of a pre-procedure screening of the patient's bone-marrow characteristics

Exclusion Criteria:

• Other cardiac or vascular system or other health-related criteria which may be seen in a patient's history and physical examination.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2025-02 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
A composite endpoint based on a 3-tiered Finkelstein-Schoenfeld (FS) hierarchical analysis. | 12 Months
  The tiers include (1) all-cause death, (2) non-fatal MACCE events, and (3) change for 6MWD from baseline to month 12.

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 12 months
  Mean change in quality of life score as measured by the MLHFQ at 12 months compared to baseline (superiority, treatment vs sham)
Survival | 12 Months
  Overall survival compared between both study arms (non-inferiority, treatment vs sham)
Time to first Major Adverse Cardiac Events (MACE) | 12 months
  Time to first MACE, defined as the composite of all-cause death, hospitalization for worsening heart failure, nonfatal recurrent myocardial infarction, placement of a left ventricular assist device (LVAD), or heart transplantation (non-inferiority, treatment vs sham)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Pepine, MD, Principal Investigator — University of Florida; Amish Raval, MD, Principal Investigator — University of Wisconsin, Madison; Duncan Stewart, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (24):
- United States (20):
  - Mayo Clinic, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford Medical Center, Stanford Health Care, Palo Alto, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado, Denver, Aurora, Colorado
  - Morton Plant Mease Health Care, Clearwater, Florida
  - University of Florida - College of Medicine/ div of Cardiovascular Medicine, Gainesville, Florida
  - Iowa Heart, Des Moines, Iowa
  - John Hopkins University School of Medicine - Dept of Cardiology, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Michigan Heart - St.Joseph Mercy Health System (Trinity Health), Ypsilanti, Michigan
  - Atlantic Health System, Morristown, New Jersey
  - New York University School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Heart, Tulsa, Oklahoma
  - Stern Cardiovascular Foundation, Memphis, Tennessee
  - Virginia Commonwealth University (VCU) Medical Center, Richmond, Virginia
  - Division of Cardiovascular Medicine, University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (4):
  - St. Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences Center, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Unity Health Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raval AN, Johnston PV, Duckers HJ, Cook TD, Traverse JH, Altman PA, Dhingra R, Hematti P, Borrello I, Anderson RD, Pepine CJ. Point of care, bone marrow mononuclear cell therapy in ischemic heart failure patients personalized for cell potency: 12-month feasibility results from CardiAMP heart failure roll-in cohort. Int J Cardiol. 2021 Mar 1;326:131-138. doi: 10.1016/j.ijcard.2020.10.043. Epub 2020 Oct 20. PMID 33091520
- [Derived] Raval AN, Cook TD, Duckers HJ, Johnston PV, Traverse JH, Abraham WT, Altman PA, Pepine CJ. The CardiAMP Heart Failure trial: A randomized controlled pivotal trial of high-dose autologous bone marrow mononuclear cells using the CardiAMP cell therapy system in patients with post-myocardial infarction heart failure: Trial rationale and study design. Am Heart J. 2018 Jul;201:141-148. doi: 10.1016/j.ahj.2018.03.016. Epub 2018 Apr 3. PMID 29803986
- See also: Website for the study sponsor — http://www.biocardia.com